CLINICAL TRIAL: NCT02062359
Title: Phase II Study of CD62L+-Derived T Lymphocytes Transduced With a T Cell Receptor Recognizing the NY-ESO-1 Antigen and Aldesleukin Following Lymphodepletion in Patients With NY-ESO-1 Expressing Melanoma
Brief Title: T Cell Receptor Immunotherapy Targeting NY-ESO-1 for Patients With NY-ESO-1 Expressing Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed due to poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140058; 14-C-0058
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Cancer; Metastatic Melanoma
Keywords: Malignant Melanoma; Metastatic Cancer; Gene Therapy; Immunotherapy; Tumor Regression
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma | interventions — Antigens, Differentiation; aldesleukin; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): Patients will receive the standard National Cancer Institute (NCI) Surgery Branch non-myeloablative, lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous (IV) infusion of the anti-NY ESO-1 T cell receptor (TCR) cluster of differentiation 62L (CD62L)+ engineered peripheral blood lymphocyte (PBL) and aldesleukin
  Interventions: Biological: Anti-NY ESO-1 T cell receptor (TCR) cluster of differentiation 62L (CD62L)+ cells; Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Anti-NY ESO-1 T cell receptor (TCR) cluster of differentiation 62L (CD62L)+ cells — Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-NY ESO-1 T cell receptor (TCR) CD62L+ cells and high dose aldesleukin.
  On day 0, cells (1x10e9 to 2x10e11) will be infused intravenously on the Patient Care Unit over 20-30 minutes.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes approximately every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
Drug: Cyclophosphamide — On days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
Drug: Fludarabine — On days -5 to -1: Fludarabine 25 mg/m(2)/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with melanoma that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying them, and then giving the cells back to the patient. In a previous study, the NCI Surgery Branch used the anti-ESO-1 gene and a type of virus (retrovirus) to make these tumor-fighting cells (anti-ESO-1 cells). About half of the patients who received this treatment experienced shrinking of their tumors. In this study, we are using a slightly different method of producing the anti-ESO-1 cells selected for a specific cell type, which we hope, will be better in making the tumors shrink.

Objectives:

The purpose of this study is to see if these tumor fighting cells (genetically modified cells) that express the receptor for the ESO-1 molecule on their surface can cause melanoma tumors to shrink and to see if this treatment is safe.

Eligibility:

-Adults 18 and older with cancer that has the ESO-1 molecule on tumor surfaces

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti ESO-1 cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the anti-ESO 1 cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
Background:

* A T cell receptor (TCR) that recognizes the NY-ESO-1 (ESO) tumor/testes antigen has been cloned into a retrovirus and can be used to genetically modify human peripheral blood lymphocytes (PBL) so they recognize human leukocyte antigen (HLA)-A2+, ESO+ tumors
* PBL expressing the anti-ESO TCR have been administered with aldesleukin with or without ALVAC vaccine to 21 patients with melanoma following lymphodepleting chemotherapy at the Surgery Branch, resulting in objective tumor regression (complete or partial regression) in ten patients (47%).
* In animal models using murine cells and in experiments with human T cells in vitro, T cell subsets expressing the lymphoid homing and differentiation marker cluster of differentiation 62L (CD62L), including na(SqrRoot) ve T cells (TNaive), stem cell memory T cells (TSCM), and central memory T cells (TCM), were shown to have superior attributes compared to whole PBL and CD62L- PBL for adoptive cell therapy, including superior persistence following transfer in vivo.

Objectives:

Primary objective:

- To determine whether the administration of anti-ESO TCR engineered CD62L+-derived lymphocytes plus high-dose aldesleukin following a non-myeloablative lymphodepleting preparative regimen can result in an objective regression rate (partial response (PR) + complete response (CR)) of melanoma tumors.

Secondary objectives:

* Determine the persistence of genetically engineered, adoptively transferred CD62L+ derived lymphocytes.
* Determine the toxicity profile of this treatment regimen.

Eligibility:

Patients who are:

* Human leukocyte antigen (HLA)-A*0201 positive
* 18 years of age or older
* Have metastatic melanoma that expresses the ESO antigen

Patients may not have:

- Contraindications for high dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cells (PBMC) will be obtained by leukapheresis and will undergo positive selection for CD62L using a CliniMACS magnetic cell separation apparatus to enrich for the less differentiated TNaive, TSCM, and TCM subsets.
* The enriched CD62L+ lymphocytes will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth, then transduced with the anti-ESO TCR.
* All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine.
* On day 0 patients will receive anti-ESO TCR gene-transduced CD62L+ -derived lymphocytes and then begin high dose aldesleukin.
* A complete evaluation of evaluable lesions will be conducted 6 weeks (+/- 2 weeks) following the administration of the cell product.
* The primary objective will be efficacy. The study will be conducted using a phase II optimal design (Simon R, Controlled Clinical Trials 10:1-10, 1989) in order to rule out an unacceptably low 40% overall response rate (p0=0.40) in favor of an improved response rate of 65% (p1=0.65). This study will initially enroll 11 evaluable patients, and if 0 to 5 of the 11 have a response, then no further patients will be accrued. If 6 or more of the first 11 patients have a response, then accrual would continue until a total of 20 patients have been enrolled. If there were 11 or more responses in 20 patients (55%), this would be sufficiently interesting to warrant further study in later trials. To allow for a very small number of inevaluable patients, the accrual ceiling will be set at 22 patients.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma that expresses ESO as assessed by one of the following methods: reverse transcription-polymerase chain reaction (RT-PCR) on tumor tissue, or by immunohistochemistry of resected tissue, or serum antibody reactive with ESO.
2. Confirmation of diagnosis of metastatic melanoma by the Laboratory of Pathology of the National Cancer Institute (NCI).
3. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
4. Greater than or equal to 18 years of age and less than or equal to 70 years of age.
5. Willing to sign a durable power of attorney
6. Able to understand and sign the Informed Consent Document
7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1
8. Life expectancy of greater than three months
9. Patients must be human leukocyte antigen (HLA)-A*0201 positive
10. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment
11. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
12. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
13. Hematology

    * Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim
    * White blood cell (WBC) greater than or equal to 3000/mm(3)
    * Platelet count greater than or equal 100,000/mm(3)
    * Hemoglobin > 8.0 g/dl
14. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal
    * Serum creatinine less than or equal to 1.6 mg/dl
    * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dl.
15. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

    Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in Section 2.1.
16. Six weeks must have elapsed from the time of any antibody therapy that could affect an anti cancer immune response, including anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody therapy, toat the time the patient receives the preparative regimen to allow antibody levels to decline.

Note: Patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
3. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms
8. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45%. Testing is required in patients with:

   * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   * Age greater than or equal to 60 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg SA, Yang JC, Sherry RM, Kammula US, Hughes MS, Phan GQ, Citrin DE, Restifo NP, Robbins PF, Wunderlich JR, Morton KE, Laurencot CM, Steinberg SM, White DE, Dudley ME. Durable complete responses in heavily pretreated patients with metastatic melanoma using T-cell transfer immunotherapy. Clin Cancer Res. 2011 Jul 1;17(13):4550-7. doi: 10.1158/1078-0432.CCR-11-0116. Epub 2011 Apr 15. PMID 21498393
- [Background] Dudley ME, Yang JC, Sherry R, Hughes MS, Royal R, Kammula U, Robbins PF, Huang J, Citrin DE, Leitman SF, Wunderlich J, Restifo NP, Thomasian A, Downey SG, Smith FO, Klapper J, Morton K, Laurencot C, White DE, Rosenberg SA. Adoptive cell therapy for patients with metastatic melanoma: evaluation of intensive myeloablative chemoradiation preparative regimens. J Clin Oncol. 2008 Nov 10;26(32):5233-9. doi: 10.1200/JCO.2008.16.5449. Epub 2008 Sep 22. PMID 18809613
- [Background] Klebanoff CA, Gattinoni L, Torabi-Parizi P, Kerstann K, Cardones AR, Finkelstein SE, Palmer DC, Antony PA, Hwang ST, Rosenberg SA, Waldmann TA, Restifo NP. Central memory self/tumor-reactive CD8+ T cells confer superior antitumor immunity compared with effector memory T cells. Proc Natl Acad Sci U S A. 2005 Jul 5;102(27):9571-6. doi: 10.1073/pnas.0503726102. Epub 2005 Jun 24. PMID 15980149
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0058.html

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Patients will receive the standard NCI Surgery Branch non-myeloablative, lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by IV infusion of the anti-NY ESO-1 TCR CD62L+ engineered PBL and aldesleukin Anti-NY ESO-1 TCR CD62L+ cells: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-NY ESO-1 TCR CD62L+ cells and high dose aldesleukin.
  On day 0,cells (1x10e9 to 2x10e11) will be infused intravenously on the Patient Care Unit over 20-30 minutes.
  Aldesleukin: Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
  Cyclophosphamide: On days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: On days
Period: Overall Study
Arm/Group | All Participants
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Response (CR) + Partial Response (PR)) of Melanoma Tumors
Description: Response was determined by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progression (PD) is at least a 20% increase in the sum of the LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 3 months
Population: None of the participants achieved a complete response or partial response and no data were collected for this assessment.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Persistence of Genetically Engineered, Adoptively Transferred Cluster of Differentiation 62L (CD62L) + Derived Lymphocytes
Description: Estimate the persistence of cells via enzyme linked immunosorbent spot (ELISPOT) and tetramer analysis by fluorescence activated cell sorting (FACS).
Time Frame: 3 months
Population: No data was collected or analyzed, thus we did not perform an evaluation of persistence for this trial. The reason is that we did not accrue a sufficient number of patients in a timely manner. A minimum of 22 subjects was needed to perform an analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2)
Hypotension (Cardiac disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Blood infection (Infections and infestations) | 1 (1)
Decreased hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Decreased platelet count (Blood and lymphatic system disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was closed due to poor accrual and the lower than expected expression of NY-ESO in participants screened.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No